CLINICAL TRIAL: NCT02265757
Title: Comparative Effectiveness of Behavioral Interventions to Prevent or Delay Dementia (CEBIPODD)
Brief Title: Behavioral Interventions to Prevent or Delay Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Julie A. Fields, Ph.D., L.P., PI, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-000885
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Mild Cognitive Impairment; Memory Disorders; Mild Dementia; Impaired Cognition; Mild Cognitive Disorder; Amnestic Disorder; Dementia and Amnestic Conditions; Poor Short-term Memory; Memory Impairment
Keywords: Behavioral Intervention; Mild Cognitive Impairment; HABIT; Cognitive Rehabilitation; Multi-Component Intervention
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Cognition Disorders; Neurocognitive Disorders; Dementia; Habits | interventions — Cognitive Training; Self-Help Groups; Exercise; Yoga

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- No Cognitive Rehabilitation (Experimental): Will receive a 10 day intervention program (over 2 weeks) consisting of Computer Brain Fitness Training, Support Group, Wellness Education and Physical Exercise.
  Interventions: Behavioral: Computer Brain Fitness Training; Behavioral: Support Group (patient and partner); Behavioral: Wellness Education; Behavioral: Physical Exercise
- No Computer Brain Fitness Training (Experimental): Will receive a 10 day intervention program (over 2 weeks) consisting of Cognitive Rehabilitation, Support Group, Wellness Education and Physical Exercise
  Interventions: Behavioral: Cognitive Rehabilitation; Behavioral: Support Group (patient and partner); Behavioral: Wellness Education; Behavioral: Physical Exercise
- No Support Group (Experimental): Will receive a 10 day intervention program (over 2 weeks) consisting of Cognitive Rehabilitation, Computer Brain Fitness Training, Wellness Education and Physical Exercise
  Interventions: Behavioral: Cognitive Rehabilitation; Behavioral: Computer Brain Fitness Training; Behavioral: Wellness Education; Behavioral: Physical Exercise
- No Wellness Education (Experimental): Will receive a 10 day intervention program (over 2 weeks) consisting of Cognitive Rehabilitation, Computer Brain Fitness Training, Support Group, and Physical Exercise
  Interventions: Behavioral: Cognitive Rehabilitation; Behavioral: Computer Brain Fitness Training; Behavioral: Support Group (patient and partner); Behavioral: Physical Exercise
- No Physical Exercise (Experimental): Will receive a 10 day intervention program (over 2 weeks) consisting of Cognitive Rehabilitation, Computer Brain Fitness Training, Support Group, and Wellness Education
  Interventions: Behavioral: Cognitive Rehabilitation; Behavioral: Computer Brain Fitness Training; Behavioral: Support Group (patient and partner); Behavioral: Wellness Education

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — Will provide each couple with memory compensation training 5 days per week for 2 weeks, with initial and ending adherence sessions. All sessions will involve 45- 60 minutes of training. The curriculum is described briefly here.
  Learning phases. three training stages from learning theory: 1) an acquisition phase in which use of the memory compensation system is learned, 2) an application phase in which a participant is taught to apply to his/her daily life, and 3) an adaptation phase in which a participant practices incorporating into his/her daily life so as to make its use habitual.
  Other Names: Memory Compensation Training; Memory Support System
  Arms: No Computer Brain Fitness Training; No Physical Exercise; No Support Group; No Wellness Education
Behavioral: Computer Brain Fitness Training — Will use the commercially available Posit Science product BrainHQ™ (www.brainhq.com) on tablets (e.g. iPads). Participants will complete 45-60 minutes of training daily in the program and will be encouraged to maintain 250 minutes of computerized brain training per week for 18 months post program. Each participant's adherence and progress will be tracked through the clinician portal provided by Posit Science both during HABIT and for 18 months post-program.
  Other Names: Brain Fitness
  Arms: No Cognitive Rehabilitation; No Physical Exercise; No Support Group; No Wellness Education
Behavioral: Support Group (patient and partner) — Patient: The patient support group will meet for 45-60 minutes daily. It will use the LifeBio Memory Journal© as a basis for reminiscence-focused group sessions. Partner: The care partner support group meets separately from the patient group for 45-60 minutes daily.
  Arms: No Cognitive Rehabilitation; No Computer Brain Fitness Training; No Physical Exercise; No Wellness Education
Behavioral: Wellness Education — The education component will involve daily 60-minute group sessions with topics including Introduction to the Program, Living with MCI, Changes in Roles, Communication and Relationships, Sleep Hygiene, Steps to Healthy Brain Aging, Preventing Dementia, MCI and Depression, Nutrition and Exercise, Safety and Assistive Technologies, and Participating in Research, Community Resources, Meaning and Purpose, and Joy.
  Arms: No Cognitive Rehabilitation; No Computer Brain Fitness Training; No Physical Exercise; No Support Group
Behavioral: Physical Exercise — The HABIT physical exercise intervention is intended to initiate and sustain a schedule rather than a type of physical activity. HABIT will provide a customized DVD as a supplement for continued use and practice after the program to those that opt to continue yoga. Will use an activity log completed by the partner to track activity level of the participants during the 18 month follow-up period.
  Other Names: Yoga
  Arms: No Cognitive Rehabilitation; No Computer Brain Fitness Training; No Support Group; No Wellness Education

SUMMARY:
This study will compare the effectiveness of different combinations of 5 types of behavioral interventions across patient-centered outcomes. It will also evaluate which outcomes (e.g. quality of life, cognition, function, mood) matter most to people at risk for dementia and their care partners. The results of this study have the potential to direct patients, families, and health care providers as to which combinations of behavioral interventions provide the greatest potential impact on which dementia prevention outcomes. Greater use of behavioral strategies that are targeted to the outcomes of most important to the patient will likely improve patient compliance and treatment adherence. This, in turn, can lessen the need for medication, health care, and long term care utilization.

DETAILED DESCRIPTION:
Traditional randomized controlled trials (RCTs) can be thought of as 'additive' trials where randomization leads to the addition of treatments beyond placebo. Participants are confronted with the probability of receiving placebo (no treatment). This leads many potential participants to not consent or to withdraw if they believe they are receiving no treatment. In contrast, the proposed trial will be 'subtractive'. This innovative approach to randomization will involve suppression of just 1 of the 5 treatment components. Thus, all participants will receive at least 80% of the menu of interventions offered in this trial.

ELIGIBILITY:
Inclusion Criteria:

A candidate for the HABIT program with a diagnosis of amnestic MCI (confirmed at eligibility visit by a Clinical Dementia Rating (CDR) scale of 0.5).

A cognitively normal care partner who has at least twice-weekly contact with the participant.

Either not taking or stable on memory medicine(s) (e.g. donepezil) for at least 3 months.

Fluent in English. (Expanding the program to communities of Spanish- speakers will be a high priority in subsequent dissemination work).

Exclusion Criteria:

Inclusion in another clinical trial that would exclude participation. Subject will be considered for participation at the end of such a trial or as appropriate.

Medically unable to participate in all arms by virtue of visual or auditory impairments or non-ambulatory status.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2014-06; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Improvement in patient quality of life | baseline to 18 months
  quality of life measured by the QOL-AD scale

SECONDARY OUTCOMES:
improvement in patient memory based everyday functioning | baseline to 18 months
  measured by the Everyday Cognitive Functioning scale (ECOG)
improvement in caregiver mood and sense of burden | baseline to 18 months
  measured by the Caregiver Burden questionnaire and the Center for Epidemiological Studies Depression scale (CESD)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fields, PhD, LP, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Levy SA, Smith G, De Wit L, DeFeis B, Ying G, Amofa P, Locke D, Shandera-Ochsner A, McAlister C, Phatak V, Chandler M. Behavioral Interventions in Mild Cognitive Impairment (MCI): Lessons from a Multicomponent Program. Neurotherapeutics. 2022 Jan;19(1):117-131. doi: 10.1007/s13311-022-01225-8. Epub 2022 Apr 12. PMID 35415779
- [Derived] Chandler MJ, Locke DE, Crook JE, Fields JA, Ball CT, Phatak VS, Dean PM, Morris M, Smith GE. Comparative Effectiveness of Behavioral Interventions on Quality of Life for Older Adults With Mild Cognitive Impairment: A Randomized Clinical Trial. JAMA Netw Open. 2019 May 3;2(5):e193016. doi: 10.1001/jamanetworkopen.2019.3016. PMID 31099860
- [Derived] Smith G, Chandler M, Locke DE, Fields J, Phatak V, Crook J, Hanna S, Lunde A, Morris M, Graff-Radford M, Hughes CA, Lepore S, Cuc A, Caselli M, Hurst D, Wethe J, Francone A, Eilertsen J, Lucas P, Hoffman Snyder C, Kuang L, Becker M, Dean P, Diehl N, Lofquist M, Vanderhook S, Myles D, Cochran D. Behavioral Interventions to Prevent or Delay Dementia: Protocol for a Randomized Comparative Effectiveness Study. JMIR Res Protoc. 2017 Nov 27;6(11):e223. doi: 10.2196/resprot.8103. PMID 29180344

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT02265757/Prot_SAP_000.pdf